CLINICAL TRIAL: NCT00829881
Title: Betahistine: Novel Therapeutic in Attention Deficit Hyperactivity Disorder
Brief Title: Effects of Using Betahistine to Treat Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: P2D, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Charles H. Pierce, MD, PhD, CPI, P2D, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R43MH082461 (NIH); R43MH082461 (NIH); MH082461; DNBBS BT-BU
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Participants will receive a placebo capsule, administered orally, once per study visit.
  Interventions: Drug: Placebo Capsule
- 2 (Experimental): Participants will receive a betahistine capsule, administered orally, once per study visit.
  Interventions: Drug: Betahistine Hydrochloride

INTERVENTIONS:
Drug: Betahistine Hydrochloride — A single betahistine hydrochloride capsule, increasing in dose from 50 mg, to 100 mg, to 200 mg, over 3 weeks
  Arms: 2
Drug: Placebo Capsule — A single placebo capsule
  Arms: 1

SUMMARY:
This study will determine whether the drug betahistine increases focus and causes side effects in people with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a disorder in which problems with paying attention and focusing disrupt people's lives. Betahistine is a drug that activates histamine, a compound found in the human body that regulates immune response and acts as a neurotransmitter. Increased availability of histamine in the brain is known to enhance attention and cognition. In previous studies, betahistine increased vigilance in healthy participants. Presently, betahistine is used outside the United States to treat vertigo, but at doses that are too low to have an effect on attention and cognition. Based on data regarding the use of betahistine outside the United States and on data from other studies using betahistine, there do not appear to be any significant side effects from its use at low doses. This study will determine both whether betahistine is effective in increasing vigilance in people with ADHD and whether it has any side effects at higher doses.

Participation in this study will last approximately 4 weeks. Participants will first attend a screening visit that will include a review of their medical and psychiatric history, a physical examination, vital signs measurements, an electrocardiogram (EKG) test, blood and urine sample collection, an eating questionnaire, and a clinical interview to confirm an ADHD diagnosis. Eligible participants will then be randomly assigned to receive either betahistine or placebo on subsequent study visits.

Participants will then attend three weekly study visits, starting 1 week after completing screening. At each visit, participants will receive a dose of either betahistine or placebo. The dose of betahistine will increase at each visit, starting at 50 mg, then increasing to 100 mg, and then to 200 mg. Participants will be asked to refrain from eating and to drink only water in the 12 hours prior to study visits. Also at each visit, participants will have their vital signs measured, complete questionnaires concerning appetite and mood, perform attention and memory tests, provide several blood samples, undergo an EKG test, and perform a breathing test. Some of these tests will be repeated several times over the course of each study visit. Additionally, at the last study visit, participants will undergo a physical examination and provide urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of attention deficit hyperactivity disorder (ADHD), combined subtype, using DSM-IV criteria
* Otherwise healthy, as determined by medical history, physical examination, and clinical laboratory tests
* Symptomatic impairment with ADHD, as evidenced by a symptom severity score of 20 or greater on the 18-item ADHD total symptom score of the Conners Adult ADHD Rating Scales (CAARS)
* Body mass index (BMI) less than or equal to 32.4 kg/m2, with a waist circumference less than or equal to 40 inches for males

Exclusion Criteria:

* Known allergies to betahistine
* Participation in a study involving administration of an investigational compound within the past month
* Pregnant
* Positive for HIV, hepatitis B antigen, or hepatitis C antibody
* Use of illicit drugs (excluding psychostimulants for ADHD) or alcohol
* History of drug addiction or alcohol abuse requiring treatment within the past 12 months
* History of asthma, peptic ulcer disease, or pheochromocytoma
* History of any other illness or condition that, in the opinion of the principal investigator, might interfere with study participation, confound the results of the study, or pose additional risk to the subject

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Attention, measured on the Continuous Performance Test through the signal detection parameter or stimulus detectability | Measured 2 and 4 hours after dosing at each of three study visits

SECONDARY OUTCOMES:
Adverse events | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Charles H. Pierce, MD, PhD, Principal Investigator — P2D, Inc.
Locations (1):
- University of Cincinnati; Department of Psychiatry, Cincinnati, Ohio, United States